CLINICAL TRIAL: NCT06879080
Title: Maternal Iron Deficiency and Childhood Health- a Prospective Cohort Study
Brief Title: Maternal Iron Deficiency and Childhood Health
Acronym: MATILDA
Status: Recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R24005
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-10

CONDITIONS: Iron Deficiency Anaemia in Childbirth; Iron Deficiency; Iron Deficiency in Pregnancy; Iron Deficiency Anemia in Pregnancy; Iron Status
Keywords: iron deficiency, iron deficiency anemia, pregnancy, pregnancy outcomes, health of the offspring
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant women recruited to the study: All pregnant women who come for prenatal visits or for labor to Tampere University Hospital, and have given their informed consent to participate to this study, and filled the electronical questionnaire about the possible iron deficiency, iron deficiency anemia, iron supplementation, folic acid use, and possible intravenous iron infusions given in pregnancy. The exposure of interest is iron deficiency and iron supplementation therapy.
- Nested cohort 1: Once the mothers have given their consent to participate this MATILDA study, we identify 100 mothers with ID/IDA, who have used iron supplement and/or given i.v. iron infusions. They are recruited in chronological order inside the bigger cohort for this nested cohort study number 1. The iron status of the mothers will be tested before delivery, and the iron status of the newborn will be followed as described in study description.
- Nested cohort 2: Prospective recruitment for the study will be continued for 2 years, and during this period we recruit 100 mothers who have had diabetes and insulin therapy in pregnancy, to this nested cohort study 2 from Tampere University Hospital. They are recruited in chronological order inside the bigger cohort for this nested cohort study number 2. The iron status of the mothers will be tested before delivery, and the iron status of the newborn will be followed as described in study description.
- Nested cohort controls: For the nested cohort groups 1 and 2, a 100 mothers without ID/IDA/diabetes will be recruited. The same controls are used for both the nested cohort groups. They are recruited in chronological order inside the bigger cohort for this control group. The iron status of the mothers will be tested before delivery, and the iron status of the newborn will be followed as described in study description.

SUMMARY:
The aim of this prospective observational cohort study is to study maternal iron deficiency and iron deficiency anemia and the use of iron supplements in pregnancy and their impact on the health of the offspring and pregnancy outcomes.

All women coming to Tampere University Hospital for prenatal checkups and/or labor are recruited to the study. After giving their consent the mothers fill an online questionnaire about about possible maternal anemia and its diagnosis in pregnancy, iron deficiency and its diagnosis in pregnancy, maternal use of iron supplement or folic acid and it´s timing, about possible other chronic disease and their medications during pregnancy, and whether the mother has got intravenous iron infusions in pregnancy. Mothers also give their permit to use their in-and outpatient data from pregnancy until hospital discharge and to follow the health of their offspring from birth until 7 years of age from in- and outpatient records.We aim to recruit 6000 mother-child-pairs.

The health of the offspring (growth, diagnoses, medication, possible therapies, need of support at daycare or school) will be followed for the first month, then at 1,5 years, four years and seven years of age from the patient records.

In addition to the cohort study, two nested cohort studies will be performed. The aim of the nested cohort studies is to study the correlation of maternal iron status to the iron status of the child. Secondary aim is to evaluate iron biomarkers, especially reticulocyte hemoglobin, and their reliability to interpret neonatal iron status.

A 100 mothers with diagnosed iron deficiency and iron supplementation (p.o. or i.v.) in pregnancy, are recruited to Nested cohort 1. For the nested cohort 2, a 100 mothers with diabetes requiring insulin therapy in pregnancy are recruited. Tor these two cohorts, a 100 mothers without iron deficiency or diabetes will be recruited as controls. Iron status of the mother will be tested before delivery from blood sample. The iron status of the offspring will be checked from umbilical blood, at 2 days of age at the same time other lab tests are taken, at eight months and two and five years of age. In addition to the laboratory tests, parents fill up an electronical questionnaire at eight months, two and five years about the nutrition, sleep, behaviour and cognitive and motor skills of their child.

The researchers try to find out, whether iron deficiency in pregnancy has long-term effects on the health and development of the offspring, and how the iron status correlates between the mother and the child, and does it have impact on their sleep, behaviour or skills.

DETAILED DESCRIPTION:
This will be a prospective cohort study in Tampere University hospital and The Wellbeing Services County of Pirkanmaa(Pirha). All pregnant women are recruited to participate to the study once they come to Tampere University Hospital for prenatal visits, for labor and/or at newborn pediatric examination performed by pediatricians usually at 2 days of age.

After giving their online consent the mothers fill up a questionnaire online about possible maternal anemia and its diagnosis in pregnancy, iron deficiency and its diagnosis in pregnancy, maternal use of iron supplement or folic acid and it´s timing, about possible other chronic disease and their medications during pregnancy, and whether the mother has got intravenous iron infusions in pregnancy. Mothers are also asked for permission to collect their patient and medication data during pregnancy to improve the reliability and coverage or the study.

Prospective recruitment for the study will be continued for 3,5 years. We aim for approximately 6000 mother- newborn pairs, of which approximately one third (2000 mothers) have got iron supplementation in pregnancy.

The health of the offspring will be followed from inpatient records at The Wellbeing Services County of Pirkanmaa from birth until 7 years of age as described at specific aims. Information about neonatal outcomes recorded as they are recorded to the Finnish Medical Birth Registry are collected from the first 7 days of life. Neonatal health is followed also until 1 month of age or until hospital discharge from in- and outpatient records. At the next follow-up time points: 1.5 years, 4 years and 7 years of age, the information (growth, possible diagnoses, possible medications, need of support at school at 7 years of age), will be collected from the outpatient records at Health and Wellbeing Services of Pirkanmaa.

Nested cohort 1 Once the mothers have given their consent to participate this MATILDA study, we identify 100 mothers with ID/IDA, who have used iron supplement and/or given i.v. iron infusions. They are recruited in chronological order inside the cohort for this nested cohort study number 1. A 100 control mothers without IDA/ID or diabetes, will be recruited in chronological order as well. Mothers for this nested cohort will be recruited at prenatal visits at Tampere University Hospital obstetric policlinic.

Nested cohort 2 Prospective recruitment for the study will be continued for 2 years, and during this period we recruit 100 mothers who have had diabetes and insulin therapy in pregnancy, to this nested cohort study 2 from Tampere University Hospital. For these mothers with diabetes and insulin therapy, a 100 control mothers without maternal diabetes and iron deficiency, will be recruited. The controls are the same patients in both nested cohorts. The study participants will be recruited in chronological order from prenatal hospital visits or once they come to the hospital for labor.

Mother´s hemoglobin, iron status (including reticulocyte hemoglobin) and C-reactive protein (CRP), will be tested once setting an i.v. route once they come to the hospital for delivery. The iron status of the newborn (small blood count, ferritin, transferrin receptor, reticulocytes including reticulocyte hemoglobin) and CRP, will be tested from umbilical cord blood. At 2-5 days of age at the same time once they are tested for metabolic screening or taken other laboratory tests, a small blood count and reticulocytes are being controlled. The iron status of the offspring (small blood count, ferritin, transferrin receptor, reticulocytes including reticulocyte hemoglobin) and CRP will also be controlled at 8 months, 2 years and 5 years of age.

At 8 months, 2 and 5 years, the family will be sent an electronical questionnaire with questions about the child´s diet, sleep patterns, cognitive development and behavior. The families will be reminded about the laboratory tests and questionnaires once via text message.

All the data will be stored at Tampere University Hospital´s safe research environment (Lokero) and pseudonymized before analysis. The data will be statistically analyzed in the safe research environment. The results of this study will be published in peer-reviewed international science journals. The study registry data will be held for five years after the study has ended and then destroyed following the instructions by Pirha.

Timetable Research permits and approval for this project have been received from Wellbeing Services County of Pirkanmaa and ethical committee in January 2024. The amendment for the extension of follow-up and follow-up questionnaires is brought to the ethical committee in October 2024.

Valtion tutkimusrahasto (VTR) has funded MATILDA-study in 2024. Additional funding for the nested cohorts will be applied during years 2024 and 2025 at least from Päivikki ja Sakari Sohlbergin Säätiö, Juho Vainion Säätiö, Pirkanmaan kulttuurirahasto, Lastentautien Tutkimussäätiö, Lääketieteen säätiö and Tays Tutkimussäätiö.

The data collection for this MATILDA- project has begun in April 2024. A systematic literature review for maternal iron deficiency and it´s effect in offspring health is prepared during data collection as a part of PhD project for medical student Inna Anttila. Data collection with questionnaires will last up to 3.5 years and it will be finished by the end of year 2027 the latest. The recruitment for the nested cohort studies will begin as soon as the funding has been secured, and end as soon ad 100 participants for each group 1 and 2 and 100 controls have been recruited, by the end of year 2027 the latest.

Main researcher (PI) in this MATILDA- project will be pediatrician Laura Seppälä from Tampere University Hospital (MD, PhD, neonatology fellow) and the nested cohorts will be run together with Pauliina Rinta-Jaskari (MD, pediatrician, PhD student). Other researchers in this project will be gynecologist Elli Toivonen from Tampere University hospital (MD, PhD), associate professor of developmental psychology Kati Heinonen-Tuomaala(PhD, adjunct professor), PhD student Inna Anttila (medical student) and PhD student Pilvi Saltiola (MD, GP), and perinatologist Kati Tihtonen (MD, PhD, Adjunct professor) and pediatrician Sauli Palmu (MD, PhD, acting professor).

Based on the previous studies, we assume that the incidence of iron deficiency anemia is 40% in our pregnant population, and that 38% of the mothers benefit from iron supplementation. Our assumption is that 67% of the children benefit from the maternal iron supplementation. Based on these assumptions, our power of 6000 mother-child-pairs will be suitable for several multivariable statistics and analyses (Fisher´s exact p<0.00001).

In the two nested cohorts, we use the same assumptions as in this bigger cohort. Needed samples size to study maternal iron status, iron supplementation and their impact on the iron status on the offspring is 200 mother-child units (Fisher´s exact p<0.00001). With this power calculation we assume the sample size to be sufficient also for multivariable analyses.

The results of this wide prospective study will be published in peer-reviewed international scientific journals. The results of this study can be widely used in pregnancy planning and follow up, and possibly bringnew knowledge for guidelines for iron deficiency therapy, or the diagnosis for iron deficiency in children, especially newborns.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Can read and write Finnish, Swedish or English

Exclusion Criteria:

* Illiterate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study is about maternal iron deficiency and iron deficicency anemia in pregnancy. People whose biological sex is female are eligible for this study.
Study Population: Study population consist of mothers who come for delivery to Tampere University Hospital between Apr 2024 and Dec 2027, and who have given their consent to participate to the study, and their offspring. We aim for 6000 mother-child pairs.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Health of the offspring | From birth to 7 years of age
  Information about neonatal outcomes recorded as they are recorded to the Finnish Medical Birth Registry are collected from the first 7 days of life. Neonatal health is followed also until 1 month of age or until hospital discharge from in- and outpatient records. At the next follow-up time points: 1.5 years, 4 years and 7 years of age, the information (growth, possible diagnoses, possible medications, need of support at school at 7 years of age), will be collected from the outpatient records at Wellbeing Services County of Pirkanmaa.

SECONDARY OUTCOMES:
Maternal pregnancy outcomes | From pregnancy to the end of postpartum period.
  Maternal pregnancy complications, delivery type, needed procedures and prescriptions are collected from inpatient records and analysed as maternal pregnancy outcomes.
Iron status of the newborn and it´s impact on the wellbeing of the child | From birth until 5 years of age
  Mother´s iron status (including reticulocyte hemoglobin) and C-reactive protein (CRP), will be tested once setting an i.v. route once they come to the hospital for delivery. The iron status of the newborn (small blood count, ferritin, transferrin receptor, reticulocytes including reticulocyte hemoglobin) and CRP, will be tested from umbilical cord blood. At 2-5 days of age at the same time once they are tested for metabolic screening or taken other laboratory tests, a small blood count and reticulocytes are being controlled. The iron status of the offspring (small blood count, ferritin, transferrin receptor, reticulocytes including reticulocyte hemoglobin) and CRP will also be controlled at 8 months, 2 years and 5 years of age.
  At 8 months, 2 and 5 years, the family will be sent an electronical questionnaire with questions about the child´s diet, sleep patterns, cognitive development and behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
Due to GDPR statement it is not possible to share individual patient data.